CLINICAL TRIAL: NCT05496582
Title: The Association of Transgelin-2, Metallothionein-2 and Ezrin With Asthma: A Case-control Study
Brief Title: The Association of Transgelin-2, Metallothionein-2 and Ezrin With Asthma
Status: Recruiting | Type: Observational
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Xiangya Hospital of Central South University (Other); National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHUTCM-0806
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole blood and induced sputum samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asthma: Previously disgnosed asthma patients
  Interventions: Diagnostic Test: No intervention
- Control: Healthy participants
  Interventions: Diagnostic Test: No intervention

INTERVENTIONS:
Diagnostic Test: No intervention — No intervention

SUMMARY:
Asthma is one of the most common chronic respiratory diseases. Previous study found a series of differentially expressed genes and proteins (transgelin-2, metallothionein-2, ezrin) in asthmatic rat. The aim of the study is to investigate the changes and associations of these gene with asthma in human.

DETAILED DESCRIPTION:
This study will investigate the changes and associations in asthma. In this project, the investigators will explore the changes of gene expression of transgelin-2, metallothionein-2 and ezrin in asthma and investigate their correlation with current diagnosis markers of asthma, including pulmonary function, fractional exhaled nitric oxide,eosinophil counts,immunoglobulin E, interleukin-5, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, aged 14-75 years;
2. Patients with a definite diagnosis of bronchial asthma;
3. The diagnosis of asthma according to the Global Initiative for Asthma (GINA), with positive bronchodilator responsiveness (reversibility) test;
4. Healthy volunteers without respiratory symptoms such as cough, wheezing, chest tightness or dyspnea;
5. Agree with all procedures in this trial by signing a written informed consent form.

Exclusion Criteria:

1. Patients with chronic obstructive pulmonary disease or other airway disease;
2. Complicated with other severe primary diseases (including hypertension, cancer, hyperthyroidism, bronchiectasia, cardiac insufficiency) and conditions that would prevent participation in the trial or put the participant at risk;
3. Women who are known to be pregnant or breastfeeding;
4. Not willing to participate;
5. Psychiatric history and neurological disorders can not work normally;
6. Other conditions that the researcher considers inappropriate to participate in this study.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants with asthma or non-asthma
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Difference in gene expression of transgelin-2, metallothionein-2 and ezrin between controls and asthmatic patients | Two year
  PCR test of gene expression of transgelin-2, metallothionein-2 and ezrin between controls and asthmatic patients
Association of transgelin-2, metallothionein-2 and ezrin with asthma | Two year
  Correlation analysis between gene expressions of transgelin-2, metallothionein-2, ezrin and current asthmatic tests (pulmonary function, fractional exhaled nitric oxide,immunoglobulin E, serum eosinophil counts, interleukin-5, etc)

CONTACTS AND LOCATIONS:
Overall Officials: Lei-Miao Yin, MD, Study Chair — Yueyang Hospital, Shanghai University of Traditional Chinese medicine; Jun-Tao Feng, MD, Study Director — Xiangya Hospital of Central South University
Locations (2):
- China (2):
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - Yueyang Hospital, Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided